CLINICAL TRIAL: NCT04021537
Title: Transcutaneous Vagal Nerve Stimulation Improvement of Sleep Quality in Veterans With PTSD With or Without History of Mild TBI
Brief Title: Non-invasive Nerve Stimulation and Sleep
Acronym: NINS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: N3140-R; 1RX003140A (Other Grant/Funding Number: Dept of Veterans Affairs)
Record Dates: First submitted 2019-06-25; First posted 2019-07-16 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The study is a cross-over design comparing two stimulation types. The order of stimulation is randomly assigned.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- non-invasive nerve stimulation a (Experimental): Electrical stimulation will be delivered to a location at the ear.
  Interventions: Device: non-invasive nerve stimulation
- non-invasive nerve stimulation b (Sham Comparator): Electrical stimulation will be delivered to a location at the ear for two minutes and rolled off to zero slowly.
  Interventions: Device: non-invasive nerve stimulation

INTERVENTIONS:
Device: non-invasive nerve stimulation — Electrical stimulation will be provided via a TENS unit.

SUMMARY:
People often have difficulty sleeping. Reasons are many. But, difficulty falling and staying asleep are common issues. Sleep difficulties are common in disorders such as Post Traumatic Stress Disorder. Current treatments for sleep difficulties are not effective for everyone. Better treatments are needed. In this study, the investigators are testing two nerve stimulation locations that may impact brain function in such a way that sleep is improved.

DETAILED DESCRIPTION:
People often have difficulty sleeping. Reasons are many. But, difficulty falling and staying asleep are common issues. Sleep difficulties are common in disorders such as Post Traumatic Stress Disorder. Current treatments for sleep difficulties are not effective for everyone. Better treatments are needed. In this study, the investigators are testing two nerve stimulation locations that may impact brain function in such a way that sleep is improved.

Prior to the cross-over study described here, a dosing study will be completed. Twenty Veterans with PTSD with or without history of mTBI, assessed for inclusion and exclusion per protocol, will be evaluated over three polysomnography nights with at least a one week washout period. Pseudo-randomly distributed across the three nights, each participant will be tested on three of the 10 parameters, creating a total of 60 testing sessions (6 for each parameter setting with each represented twice in each night slot). primary sleep architecture variables (slow wave sleep time, REM sleep time) and autonomic responses will be used as outcomes. The optimal dose will be selected and the study will proceed to the cross-over design phase.

ELIGIBILITY:
Inclusion Criteria:

* Condition: Hx VA/DOD criteria PTSD w or w/o mTBI and current sig symptoms of PTSD
* English fluency

Exclusion Criteria:

* Neurological injuries or conditions aside from mTBI that may affect outcome variables and/or other variables in the study
* Psychiatric issues that are unlikely to be related to trauma that may affect outcomes and/or other variables in the

  * e.g., schizophrenia
* Untreated sleep apnea

  * CPAP controlled sleep apnea is okay
* Major uncorrected sensory deficit
* Current drug or alcohol abuse

  * Drug abuse within the last two months will result in exclusion or delay
  * Marijuana use or alcohol intoxication within 2 weeks of study will be acceptable
* No pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-01-30 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-29 (Estimated)

PRIMARY OUTCOMES:
Polysomnography | One night comparison
  Polysomnography measures. Slow wave sleep time. Rem sleep time.

CONTACTS AND LOCATIONS:
Overall Officials: John B. Williamson, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bottari SA, Trifilio ER, Rohl B, Wu SS, Miller-Sellers D, Waldorff I, Hadigal S, Jaffee MS, Ferri R, Lamb DG, Porges EC, Williamson JB. Optimizing transcutaneous vagus nerve stimulation parameters for sleep and autonomic function in veterans with posttraumatic stress disorder with or without mild traumatic brain injury. Sleep. 2025 Aug 14;48(8):zsaf152. doi: 10.1093/sleep/zsaf152. PMID 40489292